CLINICAL TRIAL: NCT06694675
Title: An Observational Study on the Effect of Sevoflurane on Airway Hyperreactivity in Children with RSV Infection During the Perioperative Period.
Brief Title: The Effect of Sevoflurane on Airway Hyperreactivity During the Perioperative Period.
Status: Completed | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Liu Weiwei, associate professor of anesthesiology department, First Hospital of China Medical University
Other Study IDs: FirstHCMU-sevoflurane
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: RSV Infection in Children Less Than 5 Years of Age; General Anesthesia
Keywords: Sevoflurane; general anesthesia; RSV infection; pediatric patients
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tracheal secretions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: The nasopharyngeal swab test for RSV antigen was negative for patients with no history of respiratory infection in the past six weeks before surgery.
  Interventions: Drug: Sevoflurane (Volatile Anesthetic); Drug: propofol
- RSV group: The nasopharyngeal swab of the RSV antigen test is positive.
  Interventions: Drug: Sevoflurane (Volatile Anesthetic); Drug: propofol

INTERVENTIONS:
Drug: Sevoflurane (Volatile Anesthetic) — Sevoflurane 1%~3.5%
Drug: propofol — Propofol 9~15mg/kg/h

SUMMARY:
To investigate the effects of sevoflurane on respiratory parameters and respiratory inflammation in healthy and RSV-infected under general anesthesia and to propose suitable perioperative airway protection measures for children with respiratory virus infection undergoing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily joined this study and signed an informed consent form；
2. Age: 2-5 years old；
3. The patient should have a good general condition and no serious internal medicine comorbidities (ASA classification of the American Anesthesiology Association is Grade I); BMI ≤ 20;
4. Plan to undergo elective adenoidectomy or adenotonsillectomy with tracheal intubation.

Exclusion Criteria:

1. Children with a history of allergic asthma;
2. Children with space-occupying lesions of the chest and lungs, or acute bronchiolitis or pneumonia;
3. Children with cardiovascular diseases that may cause cough, wheezing, and other symptoms;
4. Children who used leukotriene modulators, β2 receptor agonists, anticholinergics, theophyllines, or hormonal treatment drugs within two weeks;
5. Children allergic to propofol, sevoflurane, or other anesthetic agents;
6. Children with a family history of malignant hyperthermia;
7. Children with liver and kidney dysfunction;
8. The result of rapid antigen detection and nucleic acid test for RSV was inconsistent, or children combined with pathogen infections other than RSV;
9. Children with fever.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 80
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Intraoperative ventilator parameters | After induction of general anesthesia and intubation; at the end of anesthesia
  Airway pressure(including Paw, PIP, Pplat), and pulmonary compliance.

SECONDARY OUTCOMES:
Inflammation response indications | After induction of general anesthesia and intubation; at the end of anesthesia
  The level of NLRP3 and IL-1β measured by ELISA in the tracheal secretions of the patients

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First hospital of China Mdical University, Shenyang, Liaoning
  - First Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No